CLINICAL TRIAL: NCT01167998
Title: Early Diagnosis of Malignant Melanoma Transformation in Pigmentary Skin Lesions
Brief Title: Early Diagnosis of Malignant Transformation of Pigmentary Skin Lesions
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Other Study IDs: orlucent-HMO-CTIL
Record Dates: First submitted 2010-07-21; First posted 2010-07-22 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2017-02

CONDITIONS: Malignant Melanoma; Pigmented Nevi; Skin Neoplasm
MeSH Terms: conditions — Melanoma; Nevus, Pigmented; Skin Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Malignant Melanoma is a deadly skin cancer that can be cured if diagnosed early. To date atypical pigmented skin lesions are diagnosed by appearance alone and many moles and lesions are excised unnecessarily and on the other hand malignant lesions are missed and diagnosed too late. In this study a protein conjugated to a florescent dye is spread on a suspicious pigmented lesion, the hypothesis is that this protein binds to malignant cells only and thus with a special camera that picks up the dye we can find pigmented lesions with early malignant transformation.

ELIGIBILITY:
Inclusion Criteria:

* pigmented lesion indicated for surgical excision
* over 18 years of age

Exclusion Criteria:

* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy individuals above 18 years of age with pignented skin lesions indicated for excision
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2010-07; Primary Completion 2017-12 (Actual); Study Completion 2019-12 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- : Hadassah Medical Organization,, Jerusalem, Israel